CLINICAL TRIAL: NCT04345432
Title: Gabapentin Treatment of Postural Tachycardia Syndrome (PoTS): a Pilot Study
Brief Title: Gabapentin Treatment of Postural Tachycardia Syndrome (PoTS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Ramesh Khurana, Chief Neurology Division, Department of Medicine, Medstar Health Research Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-167
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: Consented patients are randomized into one of two groups using balanced permutations generated randomization.com. Subject numbers will be ordered and placed in individually numbered, nontransparent envelopes by an independent observer. Trial medication is administered based on the randomization scheme.
  Baseline data will be collected followed by a 7-day trial phase of either gabapentin or placebo on a gradually increasing dosing schedule. Post-trial data will be collected on day 7 followed by 1-week washout period and Week 3 crossover medication.
Who Masked: Participant, Investigator
Masking Description: As each patient is consented, the PI will go to the randomization log which is numbered 1 through 12 and record the subject's study identification number and initials and date in the next available space on the form. He will then remove the large manila envelope in sequence corresponding to the subject's randomization number on the form, open the envelope, and remove the sub-envelope labeled Week 1 Medication. He will remove the packet for Week 1 day 7 and return it to the large envelope. He will then dispense the envelope "Week 1 Medication" containing packets for days 1-6 to the subject. The large manila envelope will then be placed in the subject's study chart until the next visit on Day 7.
  The PI will provide a photocopy of the randomization log to the independent observer after each patient is randomized. Only the independent observer will have the unblinding code in the event that an emergency situation arises and the code must be broken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gabapentin (Experimental): The experiment will be divided into the following phases:
  * Baseline phase - Demographic and test data will be collected prior to dispensing trial medication using all measures listed above
  * 7 day trial phase with gradual increase of dose from 100 mg/day to 600 mg/day (300 b.i.d) on day 6 of gabapentin or placebo. A single morning dose (300 mg) will be given at the lab on day 7 followed by post-trial testing (using above measures) 1 hour after drug administration.
  * 7 day drug washout phase - no medication will be taken
  * 7 day crossover trial phase - baseline measurements will be repeated and groups will switch to gabapentin or placebo. Post-trial measurements will be taken 1 hour after a single morning dose (300 mg) on day 7.
  * Follow-up phone call - Patients will be called 8-10 days after completion of study to ensure that there have been no unexpected events.
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): The experiment will be divided into the following phases:
  * Baseline phase - Demographic and test data will be collected prior to dispensing trial medication using all measures listed above
  * 7 day trial phase with gradual increase of dose from 100 mg/day to 600 mg/day (300 b.i.d) on day 6 of gabapentin or placebo. A single morning dose (300 mg) will be given at the lab on day 7 followed by post-trial testing (using above measures) 1 hour after drug administration.
  * 7 day drug washout phase - no medication will be taken
  * 7 day crossover trial phase - baseline measurements will be repeated and groups will switch to gabapentin or placebo. Post-trial measurements will be taken 1 hour after a single morning dose (300 mg) on day 7.
  * Follow-up phone call - Patients will be called 8-10 days after completion of study to ensure that there have been no unexpected events.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Gradually increasing doses of "medication" from 100 mg on day 1 to 300 mg twice a day on day 6. On day 7, the patient received a 300-mg dose from the day 7 envelope, about two hours after a light breakfast and 1 hour before data collection. The relatively low dose and gradual titration were selected to enhance compliance and reduce adverse effects, based on a rectal mechanosensitivity study.

SUMMARY:
In this pilot study, the investigator will test the usefulness of gabapentin in treating some of the symptoms associated with POTS. Gabapentin is FDA-approved to treat epilepsy and nerve pain and works by reducing excessive activity in the nervous system. This medication has also been shown to be effective in reducing bowel discomfort in patients with irritable bowel syndrome, sleeplessness, and possibly migraine headache. The investigator has observed positive results when prescribing gabapentin off-label to alleviate photosensitivity and headaches in POTS patients. The aim of this pilot study is to better quantify what the investigator has seen and evaluate whether it merits further study in a larger group.

DETAILED DESCRIPTION:
Postural orthostatic tachycardia syndrome (POTS) is a disorder of the autonomic nervous system. The autonomic nervous system regulates major bodily functions, such as blood pressure, heart rate, body temperature and sweating. Patients with POTS experience heart palpitations, lightheadedness, and increased heart rate upon standing as well as other symptoms, such as nausea, foggy headedness or inability to concentrate, sensitivity to light, migraine headaches, and trouble sleeping that may occur even when these patients are not standing. Because many POTS symptoms are attributed to excessive activity in parts of the brain, the investigator would like to study whether some of these symptoms can be reduced with a proven seizure medication, gabapentin.

The investigator will perform several simple tests on a group of POTS patients both before and after they have been treated with this drug. The tests will include non-invasive heart rate and blood pressure monitoring during a maneuver that requires the participant to exhale in a continuous manner as if blowing up a balloon, an assessment of sensitivity to light, and completion of several questionnaires that assess sleep behavior and sensitivity to heart, bowels, and bladder. Participants will take gabapentin for one week and placebo for another week. Neither the investigator nor the participant will know beforehand whether the participant is taking gabapentin or placebo. The investigator will then compare the results of pre-trial tests to post-trial tests to determine how effective gabapentin was at alleviating symptoms. If the trial is effective, the investigator expects gabapentin to reduce palpitations, decrease sensitivity to light, and improve sleep behavior.

Risks of this study may include participants developing side-effects due to the drug. Side-effects of gabapentin may include dizziness, drowsiness, diarrhea, dry mouth, constipation, vomiting, loss of balance, allergic reaction, fatigue, and indigestion. If any side-effects occur, the investigator anticipates that they will be mild because the drug will be administered at a very low dose. Any side-effects that occur are expected to resolve quickly after stopping the medication. Furthermore, by gradually increasing the dose and restricting the trial to a relatively short period of time, the investigator will limit the risk of side-effects.

Doctors and patients alike could benefit from this study by learning about a new use for an established drug to treat several of the symptoms of POTS, thereby improving patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 60 years of age
* For women of childbearing age, no missed menstrual cycles
* Diagnosis of POTS confirmed by the PI after autonomic function tests
* Able to discontinue GABAergic drugs, beta blockers, and sleep medication for one week before study start-up and for the duration of the study
* Able to read and understand English

Exclusion Criteria:

* Men and women under 18 and over 60 years of age

  * Unable to read or understand English
  * A history of gastroparesis, renal or hepatic dysfunction, cardiac arrhythmias, eye disorders and sleep apnea

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in Acute Panic Inventory (API) | at baseline, at 1 week from baseline (upon completion of first treatment), at 2 weeks from baseline (upon completion of washout period), at 3 weeks from baseline (upon completion of second treatment)
  Acute Panic Inventory is a validated 17-item (4 psychological and 13 somatic/visceral) questionnaire. Patients rate each item on a 4-point severity scale of 0 to 3, yielding a score of 0-51. An increase in API score >13 over baseline or a total score of >20 distinguished panic subjects from controls.

SECONDARY OUTCOMES:
Change in Palpitation Awareness and Severity Response | at baseline, at 1 week from baseline (upon completion of first treatment), at 2 weeks from baseline (upon completion of washout period), at 3 weeks from baseline (upon completion of second treatment)
  In the Palpitation Awareness and Severity Response, the patient identifies one or more of the eight types of palpitations and grades their severity (1-10) immediately after the Valsalva maneuver (expiratory strain of 40 mm Hg for 15 seconds).
Change in Insomnia Severity Index | at baseline, at 1 week from baseline (upon completion of first treatment), at 2 weeks from baseline (upon completion of washout period), at 3 weeks from baseline (upon completion of second treatment)
  Insomnia Severity Index is a validated 7-item questionnaire rating severity of insomnia on a 5-point (zero to 4) scale yielding a score of 0-28, with a score of >14 indicating insomnia.
Change in Photosensitivity Index | at baseline, at 1 week from baseline (upon completion of first treatment), at 2 weeks from baseline (upon completion of washout period), at 3 weeks from baseline (upon completion of second treatment)
  The Photosensitivity Index is a 10-point visual analog of scale yielding a score of 0-10 to rate glare and pain after 30-second exposure of ophthalmoscopic light in each eye in a dimly lit room. Higher score indicates greater sensitivity to light.
Change in Somatosensory Amplification Scale (SSAS) | at baseline, at 1 week from baseline (upon completion of first treatment), at 2 weeks from baseline (upon completion of washout period), at 3 weeks from baseline (upon completion of second treatment)
  The Somatosensory Amplification Scale is a validated 5-point severity scale used to investigate the possibility of perceptual amplification of symptoms. The scale covers 10 somatic and visceral sensations to quantify symptom amplification yielding a score of 0-50, with higher score indicating greater somatosensory amplification. A score >30 may reflect a highly somatizing condition.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benarroch EE. Postural tachycardia syndrome: a heterogeneous and multifactorial disorder. Mayo Clin Proc. 2012 Dec;87(12):1214-25. doi: 10.1016/j.mayocp.2012.08.013. Epub 2012 Nov 1. PMID 23122672
- [Background] Cortez MM, Digre K, Uddin D, Hung M, Blitzer A, Bounsanga J, Voss MW, Katz BJ. Validation of a photophobia symptom impact scale. Cephalalgia. 2019 Oct;39(11):1445-1454. doi: 10.1177/0333102419845641. Epub 2019 May 22. PMID 31116567
- [Background] Dooley DJ, Taylor CP, Donevan S, Feltner D. Ca2+ channel alpha2delta ligands: novel modulators of neurotransmission. Trends Pharmacol Sci. 2007 Feb;28(2):75-82. doi: 10.1016/j.tips.2006.12.006. Epub 2007 Jan 10. PMID 17222465
- [Background] Drummond PD. A quantitative assessment of photophobia in migraine and tension headache. Headache. 1986 Oct;26(9):465-9. doi: 10.1111/j.1526-4610.1986.hed2609465.x. No abstract available. PMID 3781834
- [Background] Freeman R, Wieling W, Axelrod FB, Benditt DG, Benarroch E, Biaggioni I, Cheshire WP, Chelimsky T, Cortelli P, Gibbons CH, Goldstein DS, Hainsworth R, Hilz MJ, Jacob G, Kaufmann H, Jordan J, Lipsitz LA, Levine BD, Low PA, Mathias C, Raj SR, Robertson D, Sandroni P, Schatz I, Schondorff R, Stewart JM, van Dijk JG. Consensus statement on the definition of orthostatic hypotension, neurally mediated syncope and the postural tachycardia syndrome. Clin Auton Res. 2011 Apr;21(2):69-72. doi: 10.1007/s10286-011-0119-5. No abstract available. PMID 21431947
- [Background] Gagnon C, Belanger L, Ivers H, Morin CM. Validation of the Insomnia Severity Index in primary care. J Am Board Fam Med. 2013 Nov-Dec;26(6):701-10. doi: 10.3122/jabfm.2013.06.130064. PMID 24204066
- [Background] Khurana RK. Orthostatic intolerance and orthostatic tachycardia: a heterogeneous disorder. Clin Auton Res. 1995 Feb;5(1):12-8. doi: 10.1007/BF01845493. PMID 7780285
- [Background] Khurana RK. Experimental induction of panic-like symptoms in patients with postural tachycardia syndrome. Clin Auton Res. 2006 Dec;16(6):371-7. doi: 10.1007/s10286-006-0365-0. Epub 2006 Aug 16. PMID 16915526
- [Background] Lee KJ, Kim JH, Cho SW. Gabapentin reduces rectal mechanosensitivity and increases rectal compliance in patients with diarrhoea-predominant irritable bowel syndrome. Aliment Pharmacol Ther. 2005 Nov 15;22(10):981-8. doi: 10.1111/j.1365-2036.2005.02685.x. PMID 16268973
- [Background] Lo HS, Yang CM, Lo HG, Lee CY, Ting H, Tzang BS. Treatment effects of gabapentin for primary insomnia. Clin Neuropharmacol. 2010 Mar-Apr;33(2):84-90. doi: 10.1097/WNF.0b013e3181cda242. PMID 20124884
- [Background] Nwazue VC, Arnold AC, Raj V, Black BK, Biaggioni I, Paranjape SY, Orozco C, Dupont WD, Robertson D, Raj SR. Understanding the placebo effect in clinical trials for postural tachycardia syndrome. Clin Exp Pharmacol Physiol. 2014 May;41(5):325-30. doi: 10.1111/1440-1681.12221. PMID 24606242
- [Background] Ross AJ, Ocon AJ, Medow MS, Stewart JM. A double-blind placebo-controlled cross-over study of the vascular effects of midodrine in neuropathic compared with hyperadrenergic postural tachycardia syndrome. Clin Sci (Lond). 2014 Feb;126(4):289-96. doi: 10.1042/CS20130222. PMID 23978222
- [Background] Wells R, Elliott AD, Mahajan R, Page A, Iodice V, Sanders P, Lau DH. Efficacy of Therapies for Postural Tachycardia Syndrome: A Systematic Review and Meta-analysis. Mayo Clin Proc. 2018 Aug;93(8):1043-1053. doi: 10.1016/j.mayocp.2018.01.025. Epub 2018 Jun 21. PMID 29937049
- [Background] Zeng Y, Hu D, Yang W, Hayashinaka E, Wada Y, Watanabe Y, Zeng Q, Cui Y. A voxel-based analysis of neurobiological mechanisms in placebo analgesia in rats. Neuroimage. 2018 Sep;178:602-612. doi: 10.1016/j.neuroimage.2018.06.009. Epub 2018 Jun 5. PMID 29883731